CLINICAL TRIAL: NCT05486858
Title: Differencies in the Contraction Ratio of Diaphragm Muscle Between Low Back Pain and Asymptomatic Individuals.
Brief Title: Diaphragm Function in Low Back Pain People
Acronym: LBP_DIA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: LBP_DIA
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical
Keywords: LBP; diaphragm; MSK ultrasound
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LBP individuals: People who suffer from pain in the lower back area.
  Interventions: Other: MSK ultrasonograpy; Other: sitting Functional and Lateral Reach Test
- asymptomatic individuals: People who has no low back pain in the patient history.
  Interventions: Other: MSK ultrasonograpy; Other: sitting Functional and Lateral Reach Test

INTERVENTIONS:
Other: MSK ultrasonograpy — MSK ultrasonography was used to measure the thickness of diaphragm muscle in supine and sitting position and in a relaxed and in a contracted state.
Other: sitting Functional and Lateral Reach Test — Sitting reach tests were used to measure the stability limits of the trunk in different directions. Functional reach test is for testing the forward direction and lateral reach tests are for testing the right and the left directions.

SUMMARY:
Pathomechanism of nonspecific low back pain is not clear for the researchers yet. Our aim is to evaluate the function of one of the stabilizer muscles of the low back area. Diaphragm's postural function is evident. However, we do not understand its changes of function in low back pain. Postural function of diaphragm was screened in supine position and in sitting too in a relaxed and in a contracted state. The thickness of diaphragm was measured and contraction ratio was calculated. Additionally, the stability limits of the trunk were measured. We were curios about the differencies in contraction ratio between asymptomatic and low back pain individuals.

DETAILED DESCRIPTION:
Pathomechanism of nonspecific low back pain is not clear for the researchers yet. Our aim is to evaluate the function of one of the stabilizer muscles of the low back area. Diaphragm's postural function is evident. However, we do not understand its changes of function in low back pain. The postural function of diaphragm was screened with Zonare Zone Ultrasound System in supine position and in sitting too in a relaxed and in a contracted state. The thickness of diaphragm was measured by using an elecric caliper of the ultrasound device and the contraction ratio was calculated. Additionally, the stability limits of the trunk were measured with sitting functional reach and sitting lateral reach tests. We were curios about the differencies in contraction ratio between asymptomatic and low back pain individuals.

ELIGIBILITY:
Inclusion Criteria:

* capable to get the scene of the measurements
* age is over 18

Exclusion Criteria:

* serious neurologycal disorder, which affects the performance on the functional tests
* previous surgical intervention which has been affected the trunk
* intensive pain, which prevent the individual to perform the needed positions (supine and sitting)
* serious lung disease or breathing disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female participants, over age 18, who were participated in the study voluntarily.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2025-02-08 (Estimated)

PRIMARY OUTCOMES:
MSK ultrasonography | 20 min
  An imaging procedure that allows doctors, physiotherapist to see muscles, joints, and more. For diagnosing muscle tears/strains, nerves, and arthritis. Physical therapy or injection of medicine may be next step. Involves radiology and center for musculoskeletal care.
  In our study, the thickness of diaphragm muscle was measured in supine and sitting positions. Its contraction ratio was calculated, based on the relaxed and the contracted states of the muscle.
sitting Functional and Lateral Reach Test | 5 min
  Special functional tests for testing the stability limits of the trunk. These are measured in sitting position, with the feet on the ground and without any support. The induvidual has to lean forward/right/left directions with forward stretched arms. We calculated the distance between the start and end positions of the fingers.

SECONDARY OUTCOMES:
Visual analogue scale | 1 min
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. VAS is the most common pain scale. We ask the participants to indicate with the visual analogue scale the intensity of low back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Csongrád-Csanád, Hungary

IPD SHARING:
Plan to Share IPD: Undecided